CLINICAL TRIAL: NCT06350916
Title: An Educational Mobile Application to Improve Patient Engagement and Decrease Postoperative Opioid Consumption in Patients Enrolled in an Enhanced Recovery After Surgery (ERAS) Pathway for Colorectal Surgery
Brief Title: Application to Improve Patient Engagement and Decrease Postoperative Opioid Consumption in Patients for Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00082594; LCI-GI-CRC-SEAMLESS-2020 (Other: Atrium Health)
Record Dates: First submitted 2024-03-18; First posted 2024-04-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SeamlessMD Mobile Application: Participants enrolling in SeamlessMD will be prompted by the mobile app to electronically complete a validated quality-of-life assessment, the Quality of Recovery (QoR-15) evaluation over 30 days. Participants will also be prompted by the app to record their daily narcotic consumption via an "Opioid Tracker" page that requests participants enter the number of doses taken for each narcotic medication in the last 24 hours.
  Interventions: Behavioral: SeamlessMD® Mobile Application
- Non-App User Study Participant: Participants will receive on postoperative day one (POD1) in the hospital a one-page paper survey of the same questions prompted by the SeamlessMD app regarding completion of preoperative ERAS metrics.

INTERVENTIONS:
Behavioral: SeamlessMD® Mobile Application — Mobile cloud-based applications (apps), such as SeamlessMD®, are readily accessible on smart phones and offer an innovative strategy to encourage and track patient adherence to recommended ERAS components pre- and postoperatively.
  Groups: SeamlessMD Mobile Application

SUMMARY:
The purpose of this study is to evaluate whether patient-centered educational material delivered before and immediately after surgery can help improve outcomes for patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
To analyze the impact of implementation of patient-centered educational material delivered the SeamlessMD® mobile application on perioperative Enhanced Recovery After Surgery (ERAS) metric completion rates among patients undergoing elective colorectal surgery. This is a non-interventional, prospective feasibility study. The planned study period will encompass adult patients (>18 years) scheduled to undergo an elective colorectal surgery procedure at CMC-Main during the six-month period of December 2020 to May 2021. Patients enrolling in SeamlessMD will be prompted by the mobile app to electronically complete a validated quality-of-life assessment, the Quality of Recovery (QoR-15) evaluation, five days prior to surgery, three days postoperatively, and 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Scheduled to undergo an elective colorectal surgery procedure (for benign or malignant colon or rectal pathology) at CMC-Main by one of the 5 participating colorectal surgeons (Davis, Hill, Kasten, Salo, Squires)
* Ability to provide informed consent

Exclusion Criteria:

* Emergent, non-elective colorectal procedures
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled to undergo an elective colorectal surgery procedure at Carolinas Medical Center-Main during a six-month period (December, 2020 through May, 2021).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Perioperative ERAS metric completion rate | 30 Days Following Hospital Discharge
  Completion rate for perioperative ERAS metrics
Postoperative hospital length of stay | 30 Days Following Hospital Discharge
  Postoperative hospital length of stay
Postoperative complications | 30 Days Following Hospital Discharge
  Occurrence of postoperative complications within 30 days, classified as Clavien-Dindo Grade I-V
30-day readmission | 30 Days Following Hospital Discharge
  Readmission to any hospital facility as inpatient within 30 days of surgery

SECONDARY OUTCOMES:
Postoperative Opioid Consumption | 30 Days Following Hospital Discharge
  Postoperative opioid consumption in morphine equivalent daily doses (MEDDs) as extracted from the medical administration record (MAR) for the inpatient hospitalization period

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm H Squires, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Releasing the Individual Participant Data (IPD) is not required to meet the study objectives, and therefore is not planned to be released. Additionally, there is no plan to share data, particularly individual participant data, with anyone who is not already involved in the study.